CLINICAL TRIAL: NCT04140669
Title: Automated Myocardial Performance Index Before, During and After Fetal Surgeries Using Samsung HERA W10
Brief Title: Automated Myocardial Performance Index Using Samsung HERA W10
Status: Terminated | Type: Observational
Why Stopped: Sponsor support and funding was terminated due to pandemic
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-005189
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Twin to Twin Transfusion Syndrome; Congenital Diaphragmatic Hernia; Neural Tube Defects; Lower Urinary Tract Infection
MeSH Terms: conditions — Fetofetal Transfusion; Hernias, Diaphragmatic, Congenital; Neural Tube Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Fetal Surgery Procedures: All pregnant women with a fetus diagnosed with a fetal abnormality and planning to undergo a fetal surgical procedure will be included in this single arm of the study.
  Interventions: Device: Automated Myocardial Performance Index (MPI)

INTERVENTIONS:
Device: Automated Myocardial Performance Index (MPI) — Automated Myocardial Performance Index will be performed using Samsung HERA W10 prior too fetal surgical interventions, during surgery, and following surgery.

SUMMARY:
Researchers are using Myocardial performance index (MPI) to assess fetal cardiac function before, during, and after fetal surgery in order to gain more knowledge about fetal cardiac function in high risk pregnancies and the relationship to outcomes of fetal surgical interventions.

DETAILED DESCRIPTION:
This study will evaluate the cardiac function in fetuses with specific conditions before, during, and after fetal interventions using an automated myocardial performance index. It is hypothesized that automated MPI can used to diagnosis and predict fetal cardiac dysfunction in fetal surgeries.

Ultrasound examination, including Doppler assessment, has served an axial rule in diagnosis and management of complex maternal-fetal conditions. Sonographic findings have been indicative of prognosis and have guided intervention at particular situations including intrauterine growth restriction and fetal alloimmunization. As researchers continue to investigate various sonographic parameters that would identify fetuses at increased risk of adverse outcomes, which would warrant intervention, fetal cardiac function has substantially attracted attention as a potential predictor of fetal status; subtle cardiac dysfunction may reflect functional adaptation to fetal insult.

Myocardial performance index (MPI) is a Doppler derived sonographic tool that is used to assess global fetal cardiac function. Higher MPI values have been proven to indicate ventricular dysfunction. Several studies have adopted the use of MPI as a part of fetal echocardiography, either to study normal values among fetal population or to assess fetal cardiac dysfunction in high risk pregnancy and in response to fetal intervention. Initial results have correlated MPI to adverse outcomes particularly in the presence of maternal and fetal disorders.

Fetal surgery is a unique stressful situation in which fetal cardiac function presents a critical aspect. In part, because underlying indications are commonly associated with clinically relevant myocardial dysfunction e.g. twin-to-twin transfusion syndrome (TTTS), congenital diaphragmatic hernia (CDH), neural tube defect (NTD) and lower urinary tract obstruction (LUTO). Moreover, surgery itself may be associated with significant fetal cardiac compromise. Therefore, perioperative (before, during and after the procedures) MPI may present a predictive parameter of fetal and neonatal outcomes in these high risk surgeries.

ELIGIBILITY:
Inclusion Criteria

• Pregnant women, aged 18 years or older, with one of the following prenatal diagnoses:

* Monochorionic diamniotic twin pregnancies complicated with TTTS
* Fetuses with CDH, but no other structural or chromosomal abnormalities
* Fetuses with NTD, but no other structural or chromosomal abnormalities
* Fetuses with LUTO, but no other structural or chromosomal abnormalities
* That provide written Informed Consent and is willing to comply with protocol requirements

Exclusion Criteria

* Presence of fetal cardiac anomalies, arrhythmias, associated morbid or lethal anomalies, chromosomal abnormalities
* Pregnancy complications that are known to impact fetal and neonatal outcomes (e.g. diabetes mellitus, hypertension, autoimmune disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on current pregnancy
Study Population: Pregnant women carrying a fetus with a diagnosis of TTTS, fetal NTD, fetal CDH, or fetal LUTO, and planning to undergo a fetal surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Automated MPI can used to diagnosis and predict fetal cardiac dysfunction in fetal surgeries. | 48 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials